CLINICAL TRIAL: NCT04342065
Title: Efficacy of Pre-emptive Different Doses of Oral Pregabalin Versus Celecoxib on Sevoflurane and Analgesic Consumption in Patients Subjected for Elective Lumbar Spine Fixation Surgery: a Randomized Controlled Trial
Brief Title: Pregabalin Versus Celecoxib on Sevoflurane and Analgesic Consumption in Spine Fixation Surgery
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: South Egypt Cancer Institute (Other)
Responsible Party: Principal Investigator, Alaa Ali M. Elzohry, Lecturer of Anesthesia, ICU and Pain Relief, Clinical Research Consultants, Inc.
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Assuit University
Record Dates: First submitted 2020-04-07; First posted 2020-04-10 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Post-Operative Pain
MeSH Terms: conditions — Pain, Postoperative | interventions — Celecoxib; Pregabalin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group (G) (Active Comparator): received gabapentin 300 mg capsule 2 hours preoperative and the same dose 6 hours postoperative.
  Interventions: Drug: Pregabalin 150mg
- Group (C) (Active Comparator): received celecoxib 200 mg 2 hours preoperative and the same dose 6 hours postoperative.
  Interventions: Drug: Celecoxib capsules

INTERVENTIONS:
Drug: Celecoxib capsules — received celecoxib 200 mg 2 hours preoperative and the same dose 6 hours postoperative.
  Arms: Group (C)
Drug: Pregabalin 150mg — received Pregabalin 150mg 2 hours preoperative and the same dose 6 hours postoperative.
  Arms: Group (G)

SUMMARY:
The anti-epileptic drugs such as gabapentin and other non-steroidal anti-inflammatory drugs (NSAID) such as celecoxib were used as a part of multimodal analgesia to control such pain. Gabapentin is an anticonvulsant drug that has analgesic effect in post-herpetic neuralgia, diabetic neuropathy, and neuropathic pain. Celecoxib is one of the NSAIDs, that its analgesic effect is reported in various studies by cyclooxygenase-2 (COX-2) inhibitor.

The aim of this randomized double-blinded study was to asses and compare the efficacy of using gabapentin versus celecoxib as a part of multimodal analgesia in perioperative hemodynamic control and pain relief in patients underwent posterior approach lumbar spine disc fixation surgery.

ELIGIBILITY:
Inclusion Criteria:

* American society of anesthesiologists (ASA) I and II, aged between 21-60 years old scheduled to undergo elective posterior approach lumbar spine disc surgery

Exclusion Criteria:

* Patients with a known sensitivity to celecoxib or pregabalin, psychotic disorder or cognitive impairment, history of drug dependency or substance addiction, history of chronic medical disease, the presence of coagulation disorders or pregnancy, were excluded from the study.

Ages: 21 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-02-01 (Actual)

PRIMARY OUTCOMES:
pain control | Change from Baseline Visual Analogue Scale every 4 hours for 48 hours (0=no pain 10=most sever pain)
  Visual Analogue Scale for pain measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- South Egypt Cancer Institute, Assiut University, Arab Republic of Egypt, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No